CLINICAL TRIAL: NCT00859001
Title: A Phase II, Open-Label, Prospective, Multicenter Study to Evaluate the Efficacy and Safety of Subsequent Treatment With the Zevalin (Ibritumomab Tiuxetan) Study in Patients With Follicular Grade I-II Lymphoma After 4 Cycles of Fludarabine-Mitoxantrone-Rituximab (FMR) Therapy.
Brief Title: Study to Evaluate the Efficacy and Safety of Subsequent Treatment With the Zevalin (Ibritumomab Tiuxetan) Study in Patients With Follicular Grade I-II Lymphoma After 4 Cycles of Fludarabine-Mitoxantrone-Rituximab (FMR) Therapy
Acronym: FM+R-Z
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Bologna (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FM+R-Z
Record Dates: First submitted 2009-03-09; First posted 2009-03-10 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2009-03

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — ibritumomab tiuxetan

ARMS (1):
- FM+R (Experimental): 4 cycles of FM+R plus Zevalin
  Interventions: Drug: FM+R; Drug: Zevalin (Ibritumomab Tiuxetan)

INTERVENTIONS:
Drug: FM+R — Fludarabine-Mitoxantrone-Rituximab
Drug: Zevalin (Ibritumomab Tiuxetan)

SUMMARY:
Study phase: Phase II Investigational product, dosage, and route of administration: Ibritumomab tiuxetan (Zevalin) is composed of a murine IgG1 monoclonal antibody (ibritumomab) covalently bound to the chelating agent tiuxetan. To prepare the active therapeutic agent [90Y]-ibritumomab tiuxetan, the antibody is chelated with the β-emitter yttrium-90 chloride immediately before intravenous administration. Treatment with [90Y]-ibritumomab tiuxetan is preceded by an infusion of rituximab (Rituxan, Mabthera) in order to optimize the biodistribution of radiolabeled antibody by depleting CD20 positive B-cells. Rituximab is a chimeric human/murine IgG1 monoclonal antibody. The Zevalin study regimen is given as an infusion of rituximab 250 mg/m2 and (where biodistribution imaging or dosimetry is compulsory) 185 MBq (5mCi) of [111In]-ibritumomab tiuxetan on Day 1 followed 7 to 9 days later by a single dose of 14.8 MBq/kg (0.4 mCi/kg) of [90Y]-ibritumomab tiuxetan, maximal dose of 1184 MBq (32 mCi), preceded by 250 mg/m2 of rituximab.

Indication: stage II-IV follicular lymphoma (FL) grade I-II after 4 cycles of FMR Study objectives: Evaluation of efficacy and safety of [90Y]-ibritumomab tiuxetan, as well as assessment of quality of life Patient population: Patients with after 4 cycles of treatment with FMR Study design: Prospective, multicenter, open-label study designed to treat patients with a sequential front-line treatment represented by 4 cycles FMR plus Zevalin Duration of treatment: Four months for FMR and two treatment days one week apart followed by a 12-week safety period for Zevalin Duration of study: Estimated duration of study is 18 months Primary efficacy parameter: Overall response rate and complete response rate Secondary efficacy parameters: Overall survival, Disease-free survival, health-related quality of life.

Safety parameters: Vital signs, adverse events (AEs), hematology, blood chemistry,and immunoglobulin levels Number of study centers: 4 study centers in Italy T otal number of patients, statistical rationale provided: Expected total of 55 patients. The final sample size will be based on the number of events observed for the primary efficacy endpoint as calculated in the sequential statistical model.

Adverse events: AEs observed, mentioned upon open questioning and/or spontaneously reported will be documented.

Planned start and end of recruitment: Start of recruitment: 3rd quarter 2006. End of recruitment: 1st quarter of 2007

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed FL grade I-II according to the REAL/WHO classification (from initial diagnosis made prior to starting FMR therapy);
* FLIPI 3 or more
* Central pathology review confirming the FL grade I-II diagnosis and CD20 positivity, and no evidence/evidence with an infiltration <25% of FL in bone marrow;
* The first part of the treatment of FL must have been 4 cycles of standard FM chemotherapy (fludarabine 25 mg/m2/day on days 1 to 3 and mitoxantrone 10 mg/m2 on day 1) in combination with rituximab (375 mg/m2); Complete remission (CR), unconfirmed complete remission (CRu), partial response, and non-responder according to the International Workshop Response Criteria for NHL described by Cheson et al after four cycles of FMR. CT scans of the neck, thorax, abdomen, and pelvis and PET total body must have been performed within 3 weeks after the last dose of the last course of FMR;
* Patients 18-years-of-age or older at time of accrual;
* WHO performance status (PS) of 0 to 2 within 1 week of accrual;
* Absolute neutrophil count (ANC) more than 1.5 x 109/L within 1 week of accrual;
* Hemoglobin (Hgb) more than10 g/dL within 1 week of accrual;
* Platelets more than 150 x 109/L within 1 week of accrual.
* Written informed consent obtained according to local guidelines

Exclusion Criteria:

* Presence of any other malignancy or history of prior malignancy except non-melanoma skin tumors or stage 0 (in situ) cervical carcinoma;
* Prior radioimmunotherapy, radiation therapy, or any other NHL therapy;
* Presence of gastric, central nervous system (CNS), or testicular lymphoma at first diagnosis;
* Histological transformation of low-grade NHL;
* Known seropositivity for hepatitis C virus (HCV) or hepatitis B surface antigen (HbsAg);
* Known history of HIV infection;
* Abnormal liver function: total bilirubin > 1.5 x ULN or ALT > 2.5 x ULN within 1 week of accrual;
* Abnormal renal function: serum creatinine > 2.0 x ULN within 1 week of accrual;
* Known hypersensitivity to murine or chimeric antibodies or proteins;
* G-CSF or GM-CSF therapy within two weeks (or four weeks if pegylated) prior to screening laboratory sampling;
* Concurrent severe and/or uncontrolled medical disease (e.g., uncontrolled diabetes, congestive heart failure, myocardial infarction within 6 months of study, unstable and uncontrolled hypertension, chronic renal disease, or active uncontrolled infection) which could compromise participation in the study;
* Male and female patients of child-bearing potential unwilling to practice effective contraception during the study and unwilling or unable to continue contraception for 12 months after their last dose of study treatment;
* Female patients who are pregnant or are currently breastfeeding;
* Treatment with investigational drugs less than 4 weeks before the planned Day 1 or nonrecovery from the toxic effects of such therapy;
* Surgery less than 4 weeks before the planned Day 1 or nonrecovery from the side effects of such surgery;
* Concurrent corticosteroid use for any reason except as premedication in case of known or suspected allergies to contrast media or as premedication for potential side effects of rituximab treatment;
* Unwillingness or inability to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
disease-free survival, complete response

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto di Ematologia e Oncologia Medica Seràgnoli, Bologna, BO, Italy

REFERENCES:
- [Background] Zinzani PL, Tani M, Pulsoni A, Gobbi M, Perotti A, De Luca S, Fabbri A, Zaccaria A, Voso MT, Fattori P, Guardigni L, Ronconi S, Cabras MG, Rigacci L, De Renzo A, Marchi E, Stefoni V, Fina M, Pellegrini C, Musuraca G, Derenzini E, Pileri S, Fanti S, Piccaluga PP, Baccarani M. Fludarabine and mitoxantrone followed by yttrium-90 ibritumomab tiuxetan in previously untreated patients with follicular non-Hodgkin lymphoma trial: a phase II non-randomised trial (FLUMIZ). Lancet Oncol. 2008 Apr;9(4):352-8. doi: 10.1016/S1470-2045(08)70039-1. Epub 2008 Mar 14. PMID 18342572